CLINICAL TRIAL: NCT03224182
Title: A Randomized, Multicenter, Two-Arm, Single-Dose, Double-Blind, Placebo-CONtrolled Phase 3 Study of Intravesical Qapzola™ (Apaziquone) as a Chemotherapy Adjuvant to TransUrEthral Resection of Bladder Tumors in Patients With Low- to Intermediate-Risk Non-Muscle Invasive Bladder Cancer (CONQUER)
Brief Title: A Study of Intravesical Qapzola (Apaziquone) as a Surgical Adjuvant in Participants Undergoing Transurethral Resection of Bladder Tumor (TURBT)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Suspended development
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPI-QAP-306
Record Dates: First submitted 2017-04-14; First posted 2017-07-21 (Actual); Results first posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-08

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — apaziquone

STUDY DESIGN:
Intervention Model Description: This is a randomized, multicenter, two-arm, double-blind, placebo-controlled study of Qapzola in participants with low- to intermediate-risk NMIBC.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Qapzola (Experimental): Participants were randomized to receive a single dose of Qapzola 8 mg by intravesical administration into the bladder at 60 ± 30 minutes post transurethral resection of bladder tumor (TURBT) on Day 1 via an indwelling 100% Silicone Foley catheter and retained in the bladder for 60 ± 5 minutes.
  Interventions: Drug: Qapzola
- Placebo (Placebo Comparator): Participants were randomized to receive a single dose of Qapzole-matching placebo by intravesical administration into the bladder at 60 ± 30 minutes post TURBT on Day 1 via an indwelling 100% Silicone Foley catheter and retained in the bladder for 60 ± 5 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Qapzola — Qapzola administered by the intravesical route.
  Arms: Qapzola
Drug: Placebo — Qapzole-matching placebo administered by the intravesical route.
  Arms: Placebo

SUMMARY:
This is a randomized, multicenter, two-arm, double-blind, placebo-controlled study of Qapzola in participants with low- to intermediate-risk non-muscle invasive bladder cancer (NMIBC), assessed according to the 2016 American Urology Association (AUA) Guidelines. Specifically, only participants with the following low-to intermediate-risk tumor characteristics were included in the study.

2016 American Urological Association Stratification for Non-Muscle Invasive Bladder Cancer:

Low Risk

* Low grade solitary Ta ≤3 centimeters (cm)
* Papillary urothelial neoplasm of low malignant potential (PUNLMP)

Intermediate Risk

* Recurrence within 1 year, low-grade Ta
* Solitary low-grade Ta >3 cm
* Low-grade Ta, multifocal
* High-grade Ta, ≤3 cm (solitary tumor)

DETAILED DESCRIPTION:
In addition to other Screening assessments, participants underwent an assessment of urothelial carcinoma of the bladder via cystoscopy for clinically apparent tumor of Ta histology, including PUNLMP, although participants with strongly suspected PUNLMP at Screening or transurethral resection of bladder tumor (TURBT) were not to be enrolled in the study. The qualifying cystoscopy could be performed up to 45 days prior to signing the informed consent.

Eligible participants were randomized in a 2:1 ratio to either:

* Arm 1: One dose of 8 milligrams (mg) Qapzola
* Arm 2: One dose of placebo

Once approved for randomization, participants underwent TURBT on Day 1 and the study drug instillation occurred at 60 ± 30 minutes post-TURBT and was retained for 60 minutes (±5 minutes) in the bladder. All histology specimens were reviewed by a local pathology laboratory and all clinical treatment decisions were based on the local pathology review. Participant target disease was confirmed and efficacy analyses were performed based on the pathology results. The target study population was low- to intermediate-risk participants who had Ta histology, including PUNLMP, as confirmed by a pathology laboratory. Participants with strongly suspected PUNLMP at Screening or TURBT were not to be enrolled in the study. Participants whose tumor histology did not meet the criteria for eligibility, as confirmed by pathology (Non-Target Population), were to be followed up for safety on Day 35 (±5 days) (Safety Follow-up Visit) and were discontinued from the study. If the pathology results were delayed beyond 35 days, the Safety Follow-up Visit was to be conducted when the results were available for these participants.

Participants who had pathology-confirmed target histology did not receive additional medications to treat NMIBC during the follow-up while on the study. All target disease participants were to be followed until either a confirmed tumor recurrence, additional bladder cancer treatments, or until the End-of-Study, whichever occurred first.

The primary analysis was conducted once the required number of recurrence events were observed. A recurrence was defined as any pathologically confirmed disease of ≥Ta histology or carcinoma in situ (CIS) post-treatment. The number of events needed to perform the final primary endpoint analysis was estimated based on the recurrence rate at 24 months from previous studies. The follow-up schedule is below:

* Cystoscopic examination (all participants) and urine cytology (only participants with a Baseline diagnosis of intermediate-risk NMIBC) every 3 months (±30 days) (calculated from date of TURBT) for 2 years for tumor recurrence and progression and then every 6 months (±60 days) until either a confirmed tumor recurrence or the End-of-Study, whichever occurred first.
* If at any time during the study there was a histologically confirmed tumor recurrence, the participants discontinued from the study at that time and could then be treated per the Investigator's standard of care.

The study was to end (End-of-Study) when the required number of events for the primary endpoint analysis was accrued.

Duration of Study: The duration of the study for each participant was as follows:

* Screening Period: up to 30 days
* Treatment: Day 1
* Safety Follow-up: Day 35 (±5 days) after treatment
* Follow-up Period: No follow-up in non-Target Population. Until either a confirmed tumor recurrence or the End-of-Study, whichever occurred first in the Target Population.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have had a clinical diagnosis of low- to intermediate-risk non-muscle invasive bladder cancer according to the 2016 American Urological Association (AUA) Guidelines, except for strongly-suspected papillary urothelial neoplasm of low malignant potential (PUNLMP).
2. Participant was willing to give written informed consent and was able to adhere to dosing and visit schedules, and meet all study requirements.
3. Participant was at least 18 years of age and <90 years of age at the time Informed Consent is signed.
4. Participant was willing to practice two forms of contraception, one of which must have been a barrier method, from study entry until at least 35 days after study treatment. Participants surgically sterilized or who were postmenopausal for at least 1 year (defined as more than 12 months since last menses) did not require contraception.
5. Females of childbearing potential had a negative pregnancy test within 30 days prior to randomization. Females who were postmenopausal for at least 1 year (defined as more than 12 months since last menses) or were surgically sterilized did not require this test.

Exclusion Criteria:

1. Participant had malignancy or life-threatening systemic disease or a history of advanced, serious, life-threatening malignancy/disease within the last 5 years, except very low-risk prostate cancer.
2. Participant had used any investigational drugs, biologics (vaccines, antibodies), or devices within 30 days prior to study treatment or had plans to use any of these during the course of the study.
3. Participant had received any pelvic radiotherapy (including external beam and/or brachytherapy).
4. Participant had a history of allergy to red color food dye or any other component of Qapzola, placebo, or their diluents.
5. Participant had a surgical procedure 4 weeks prior to TURBT or had other surgical procedures performed at the time of TURBT or within 4 weeks after TURBT.
6. Participant had any unstable or uncontrolled medical condition that would make it potentially unsafe to undergo TURBT including a previous stroke or myocardial infarction within 6 months.
7. Participant had an active uncontrolled infection, including a urinary tract infection, underlying medical condition, or other serious illness that would impair the ability of the participant to receive study treatment or undergo study procedures.
8. Participant had a bleeding disorder or a screening platelet count <100×10^9/per liter (L), or required continuous anticoagulation or bridging anticoagulation during the procedure.
9. Participant had a hemoglobin value <10 grams per deciliter (g/dL) at Screening.
10. Participant had confirmed extravesical urothelial disease (upper tract and urethral including prostatic urethral).
11. Participant had history of previous bladder cancer:

    * High-Risk NMIBC as classified per the 2016 AUA Guidelines
    * Bladder cancer that was muscle invasive or positive for lymph node or distant metastasis.
12. Participant had received any previous intravesical therapy for bladder cancer- chemotherapy, immunotherapy, or previous exposure to Qapzola in the previous 3 years.
13. Participant had a tumor in the bladder diverticulum.
14. Participant had a history of interstitial cystitis.
15. Participant was pregnant or breast-feeding.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shanta Chawla, MD, Study Director — Spectrum Pharmaceuticals, Inc
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with low-to intermediate-risk non-muscle invasive bladder cancer (NMIBC) were enrolled at 34 investigative sites in the United States (US) from 04 August 2017 to 26 September 2019.
Pre-assignment Details: A total of 118 participants were randomized into the study, out of which 1 participant completed the study.
Period: Overall Study
Arm/Group | Qapzola | Placebo
Started | 81 | 37
Safety Population | 73 | 36
Completed | 0 | 1
Not Completed | 81 | 36
Not completed — Study Drug Not Instilled | 6 | 1
Not completed — Histology Other than Low- to Intermediate-Risk NMIBC | 22 | 11
Not completed — Withdrew of Consent | 4 | 2
Not completed — Investigator Decision | 3 | 1
Not completed — Sponsor Decision | 26 | 12
Not completed — Participant Refused Follow-up Procedures/Cystoscopy | 4 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Participant Had Recurrence | 11 | 5
Not completed — Death | 0 | 1
Not completed — Reason not Specified | 3 | 3
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all treated participants, classified according to the actual treatment received, regardless of random assignment.
Groups:
- Qapzola: Participants were randomized to receive a single dose of Qapzola 8 mg by intravesical administration into the bladder at 60 ± 30 minutes post TURBT on Day 1 via an indwelling 100% Silicone Foley catheter and retained in the bladder for 60 ± 5 minutes.
- Total: Total of all reporting groups
Arm/Group | Qapzola | Placebo | Total
Number analyzed (Participants) | 73 | 36 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (10.28) | 68.9 (10.16) | 67.1 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 58 | 23 | 81
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 0 | 1 | 1
  Race: Black or African American | 2 | 3 | 5
  Race: White | 71 | 31 | 102
  Race: Race-Other | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 12 | 6 | 18
  Ethnicity: Not Hispanic or Latino | 58 | 29 | 87
  Ethnicity: Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to Recurrence
Description: Time from randomization to the date of histologically confirmed recurrence of bladder cancer. A recurrence was defined as any pathologically confirmed disease of ≥Ta tumor histology or carcinoma in situ (CIS) post-treatment.
Time Frame: From randomization to date of histologically confirmed recurrence of bladder cancer (up to 2.1 years)
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Qapzola | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: 2-Year Recurrence Rate
Description: The percentage of participants with histologically confirmed recurrence of the bladder tumor at any time after randomization and on or before Year 2. A recurrence was defined as any pathologically confirmed disease of ≥Ta tumor histology or CIS post-treatment.
Time Frame: 2 years
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Qapzola | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression was defined as the time from randomization to the first disease progression. The development of T2 or greater disease was only included in the assessment of time to disease progression.
Time Frame: From randomization to first disease progression (up to 2.1 years)
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Qapzola | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Event (TEAE), Treatment-related Adverse Events, Serious Adverse Events (SAEs), TEAEs Leading to Discontinuation, TEAEs of Special Interest, and Death
Description: An AE was untoward medical occurrence in a participant who had study drug without possibility of causal relationship. TEAEs: AEs that occurred from dose of treatment until 35 days after study drug administration. Treatment-related AEs included TEAEs with relationship to study treatment (possible, probable, definite/missing). SAE was AE resulting in: death; initial/prolonged inpatient hospitalization; life-threatening; persistent or significant disability/incapacity; congenital anomaly. TEAEs of special interest were AEs of grade ≥3 dysuria and hematuria per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. Grade ≥3 hematuria included gross hematuria; transfusion, hospitalization indicated; elective endoscopy, radiologic or operative intervention indicated; limiting self-care activities of daily living (ADL), life-threatening events/death. Grade ≥3 dysuria included severe pain; pain/analgesics severely interfering with ADL and disabling.
Time Frame: Up to 2.1 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Qapzola | Placebo
Number analyzed (Participants) | 73 | 36
Participants
  TEAEs | 23 | 7
  Treatment-related AEs | 8 | 4
  SAEs | 1 | 2
  TEAEs Leading to Discontinuation | 0 | 0
  TEAE of Special Interest: Dysuria | 0 | 0
  TEAE of Special Interest: Haematuria | 0 | 1
  Death | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 2.1 years
Description: Safety Population included all treated participants, classified according to the actual treatment received, regardless of random assignment.
Arm/Group | Qapzola | Placebo
All-Cause Mortality (participants affected / at risk) | 0/73 | 1/36
Serious Adverse Events (participants affected / at risk) | 1/73 | 2/36
Other Adverse Events (participants affected / at risk) | 22/73 | 6/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Qapzola (N=73) | Placebo (N=36)
Haematuria (Renal and urinary disorders) | 0 | 1
Bladder spasm (Renal and urinary disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Qapzola (N=73) | Placebo (N=36)
Urinary tract infection (Infections and infestations) | 5 | 3
Bladder spasm (Renal and urinary disorders) | 8 | 2
Dysuria (Renal and urinary disorders) | 4 | 0
Haematuria (Renal and urinary disorders) | 6 | 1

LIMITATIONS AND CAVEATS:
The study was terminated as per Sponsor's decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-12-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT03224182/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT03224182/SAP_001.pdf